CLINICAL TRIAL: NCT01450735
Title: Evaluation of the MANOS Carpal Tunnel Release System in Patients With Carpal Tunnel Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment did not reach our intended sample size due to availability of CTR with MANOS outside of the study.
Sponsor: Thayer Intellectual Property, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THA001
Record Dates: First submitted 2011-10-06; First posted 2011-10-12 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MANOS CTR™ — The MANOS device is a carpal tunnel blade used to release the transverse carpal ligament in order to provide relief for Carpal Tunnel Syndrome.

SUMMARY:
The MANOS device is a carpal tunnel blade used to perform carpal tunnel release (CTR). CTR is indicated for the treatment of Carpal Tunnel Syndrome when conservative therapy fails. This study is being conducted to evaluate the safety and effectiveness of CTR with the MANOS device.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to undergo carpal tunnel release surgery.
* Patient has chronic Carpal Tunnel Syndrome with persistent symptoms despite non-operative treatment, or refusal of non-operative treatment, with one or more of the following: splinting, NSAIDs or corticosteroid injections.
* Carpal Tunnel Syndrome must be confirmed by positive results of Electromyography (EMG) and Nerve Conduction Velocity (NCV) tests.
* Patient is a male or non-pregnant, non-lactating female.
* Patient is 18-75 years of age, inclusive.
* Female patients of child-bearing potential, including those who have had a tubal ligation, but excluding those who have not experienced a menstrual period for at least two years, must have a negative urine pregnancy test at Screening.
* Patient must voluntarily provide written, informed consent.

Exclusion Criteria:

* Patient has a prior or current musculoskeletal or neurologic condition that limits strength, motion, or sensation in the affected hand.
* Patient has a medical condition that precludes the use of anesthetic required for surgery.
* Patient has an ipsilateral injury or other conditions affecting hand function.
* Patient has acute CTS resulting from an injury (e.g., fracture).
* Patient has had previous CTR surgery on the affected hand.
* Patient has psychiatric history, head injury or any other condition which, in the Investigator's opinion, would prevent patient from complying with post-operative hand therapy or follow-up visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Gather clinical outcome data on the safety and efficacy of the MANOS Carpal Tunnel Release System. | Baseline throughout 12 weeks post-operatively
  Clinical outcome data that will be evaluated:
  * Carpal Tunnel Syndrome Questionnaire (CTSQ)
  * Scar sensitivity
  * Hand sensation
  * Grip and pinch strength
  * Hand dexterity

SECONDARY OUTCOMES:
Safety information will be evaluated by collecting the type, frequency, severity, device, and procedure-relatedness of adverse events. | Baseline throughout 12 weeks post-operatively

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Hand Treatment Center, Hayward, California
  - Neurospine Institute Medical Group, San Francisco, California
  - William Bowen, MD Orthopedic Surgery, Willits, California